CLINICAL TRIAL: NCT04129294
Title: Exploratory Study of NS-089/NCNP-02 in Duchenne Muscular Dystrophy
Brief Title: Exploratory Study of NS-089/NCNP-02 in DMD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center of Neurology and Psychiatry, Japan (Other)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hirofumi Komaki, Director, National Center of Neurology and Psychiatry, Japan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCNP/DMT02; UMIN000038505 (Other: UMIN-CTR)
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NS-089/NCNP-02 (Experimental): NS-089/NCNP-02
  Interventions: Drug: NS-089/NCNP-02

INTERVENTIONS:
Drug: NS-089/NCNP-02 — NS-089/NCNP-02 for Infusion is packaged as 50 mg/mL with 3 mL per vial. Study dosages will be infused over a 1 hour period at the following dose levels.
  "[Part 1] NS-089/NCNP-02 is administered at dose levels 1 and 3 in Cohort 1 and at dose levels 2 and 4 in Cohort 2.
  Dose level 1: 1.62 mg/kg once weekly for 2 weeks; Dose level 2: 10 mg/kg once weekly for 2 weeks; Dose level 3: 40 mg/kg once weekly for 2 weeks; Dose level 4: 80 mg/kg once weekly for 2 weeks [Part 2] Based on the results from Part 1, two dosages are selected as study dosages in Part 2. Each selected dose are administered once a week for 24 weeks."

SUMMARY:
This study is designed to assess the safety, tolerability, efficacy and pharmacokinetics (PK) of NS-089/NCNP-02 in subjects diagnosed with Duchenne muscular dystrophy (DMD), and to determine the dosage for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* Has an out of frame deletion(s) that could be corrected by skipping exon 44 as confirmed by any of methodology at the time of visit 1. If not confirmed by any of methodology that evaluates the relative copy number of all exons (i.e. MLPA etc), must be confirmed through these techniques by the time of visit 3.
* DNA sequencing of exon 44 confirms that no DNA polymorphisms occur that could compromise duplex formation between NS-089/NCNP-02 and pre-mRNA.
* Male and >= 8 years and < 17 years of age at the time of obtaining informed consent and/or assent. Subjects aged >= 4 years and < 8 years can be enrolled according to the circumstances.
* Able to give informed consent in writing signed by parent(s) or legal guardian who is able to understand all of the study procedure requirements. If applicable, able to give informed assent in writing signed by the subject.
* Life expectancy of at least 1 year
* Able to ambulate. Non-ambulant subject can be enrolled according to the circumstances.
* Have intact muscles, which have adequate quality for biopsy. (No lacks or severe atrophy of biceps brachii or tibialis anterior muscle)
* QTc <450 msec (based on 12-lead ECGs), or <480 msec for subject with Bundle Branch Block.
* Glucocorticoid-naive patients, or patients who have used systemic glucocorticoids for at least 6 months prior to enrollment in this study with no dose changes for at least 3 months prior to enrollment.

Exclusion Criteria:

* Has participated in other pharmacological clinical trial that might recover dystrophin protein by the readthrough or the exon-skipping therapy, and/or upregulate the dystrophin-associated proteins such as utrophin.
* A forced vital capacity (FVC) < 50% of predicted.
* Continuous use of artificial respirator (except for use of NPPV while sleeping)
* A left ventricular ejection fraction (EF) < 40% or fractional shortening (FS) < 25% based on echocardiogram (ECHO).
* Surgery within the last 3 months prior to the first anticipated administration of study medication or planned for anytime between visit 1 of Part 1 and the last visit of Part 2.
* Positive hepatitis B surface antigen (HbsAg), hepatitis C antibody test (HCV), or human immunodeficiency virus (HIV) test at screening.
* Current diagnosis of any immune deficiency or autoimmune disease.
* Current diagnosis of any active or uncontrolled infection, cardiomyopathy, or liver or renal disease.
* Use of any other investigational agents and/or experimental agents within 3 months prior to the first anticipated administration of study medication.
* History of any severe drug allergy.

Ages: 4 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Adverse event and adverse drug reaction [Safety and Tolerability] | At the end of Part 2 (24 weeks treatment period and 12 weeks follow up period)
  adverse event and adverse drug reaction

SECONDARY OUTCOMES:
Expression of dystrophin protein | At the end of the treatment period (24 weeks) of Part 2
  Expression of dystrophin protein
NSAA | At the end of the treatment period (24 weeks) of Part 2
  North Star Ambulatory Assessment
TTSTAND | At the end of the treatment period (24 weeks) of Part 2
  Time to Stand Test
TTRW | At the end of the treatment period (24 weeks) of Part 2
  Time to Run/Walk 10 Meters test
6MWT and 2MWT | At the end of the treatment period (24 weeks) of Part 2
  Six-Minute Walk Test (6MWT) and Two-Minute Walk Test (2MWT)
TUG | At the end of the treatment period (24 weeks) of Part 2
  Timed Up & Go (TUG) test
PUL | At the end of the treatment period (24 weeks) of Part 2
  Performance of Upper Limb test
Detection of exon 44-skipped mRNA of dystrophin in muscle tissue | At the end of the treatment period (24 weeks) of Part 2
  Detection of exon 44-skipped mRNA of dystrophin in muscle tissue
NS-089/NCNP-02 concentration of the blood plasma | At the end of Part 2 (24 weeks treatment period and 12 weeks follow up period)
  NS-089/NCNP-02 concentration of the blood plasma
Serum Creatine kinase concentration | At the end of Part 2 (24 weeks treatment period and 12 weeks follow up period)
  Serum Creatine kinase concentration

CONTACTS AND LOCATIONS:
Overall Officials: Hirofumi Komaki, MD, PhD, Principal Investigator — National Center of Neurology and Psychiatry, Japan
Locations (1):
- National Center of Neurology and Psychiatry, Kodaira, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Komaki H, Takeshita E, Kunitake K, Ishizuka T, Shimizu-Motohashi Y, Ishiyama A, Sasaki M, Yonee C, Maruyama S, Hida E, Aoki Y. Phase 1/2 trial of brogidirsen: Dual-targeting antisense oligonucleotides for exon 44 skipping in Duchenne muscular dystrophy. Cell Rep Med. 2025 Jan 21;6(1):101901. doi: 10.1016/j.xcrm.2024.101901. Epub 2025 Jan 9. PMID 39793573
- [Derived] Ishizuka T, Komaki H, Asahina Y, Nakamura H, Motohashi N, Takeshita E, Shimizu-Motohashi Y, Ishiyama A, Yonee C, Maruyama S, Hida E, Aoki Y. Systemic administration of the antisense oligonucleotide NS-089/NCNP-02 for skipping of exon 44 in patients with Duchenne muscular dystrophy: Study protocol for a phase I/II clinical trial. Neuropsychopharmacol Rep. 2023 Jun;43(2):277-286. doi: 10.1002/npr2.12335. Epub 2023 Apr 3. PMID 37326950